CLINICAL TRIAL: NCT04846985
Title: Observational Study of Nutritional Problems in Lung and Pancreas Cancer Patients in Chemotherapy
Brief Title: Nutritional Problems in Pallative Cancer
Status: Completed | Type: Observational
Sponsor: Jens Rikardt Andersen (Other)
Collaborators: Hillerod Hospital, Denmark (Other)
Responsible Party: Sponsor-Investigator, Jens Rikardt Andersen, Associate Professor, Primary Investigator, University of Copenhagen
Organization: University of Copenhagen (Other)
Other Study IDs: H-20083532
Record Dates: First submitted 2021-04-12; First posted 2021-04-15 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Lung Cancer; Pancreatic Cancer
Keywords: Malnutrition; cancer; weight loss; lean body mass
MeSH Terms: conditions — Lung Neoplasms; Pancreatic Neoplasms; Malnutrition; Neoplasms; Weight Loss

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to investigate those nutritional problems contributing to loss of lean body mass in lung and pancreas cancer patients in chemotherapy. Furthermore to investigate alterations in taste and how they correlates with changes in following factors: nutritional intake, physical activity, appetite, food preferences, side effects, fatique and meal perception.

DETAILED DESCRIPTION:
This study will include a recruitment of 50 lung and pancreas cancer patients currently in chemotherapy. They will be observed during a period of 9-12 week, including at least 2 chemotherapy treatments. The presence and severity of the nutritional problems will be examined by observing as many different factors as possible. This includes taste alterations, weight changes, nutritional intake, physical activity, interviews and weekly questionnaires. In relation to this our primary outcome is to investigate the correlation between changes in taste and changes in nutritional intake. Secondarily the investigators want to investigate nutritional intake, physical activity, appetite, food preferences, side effects, fatique and meal perception.

ELIGIBILITY:
Inclusion Criteria:

* Lung or pancreas cancer patient
* In chemoterapy regardless of line treatment with/without combined treatment
* Legal age
* Able to speak and read in danish
* Ambulant

Exclusion Criteria:

* Inability to give consent and complete questionnaires
* Participating in clinical interventions during the periode of observation
* Allergic to milk or for any reason don't consume diary products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung and pancreas cancer patients in chemotherapy.
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2021-10-07 (Actual)

PRIMARY OUTCOMES:
To investigate the correlation between changes in taste and changes in nutritional intake | 9-12 weeks (3 treatment cycles)
  Changes in taste measured by a sensory test combined with questionnaires, and changes in nutrional intake is measured by photografies of meals

CONTACTS AND LOCATIONS:
Overall Officials: Maria Elisabeth Lendorf, MD, PhD, Principal Investigator — Hillerod Hospital, Denmark
Locations (1):
- Hillerod hospital, Denmark, Hillerød, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: No